CLINICAL TRIAL: NCT05661669
Title: Ketamine for the Treatment for Alcohol Use Disorder in the Emergency Department: A Pilot Double-blind, Placebo-controlled Randomized Clinical Trial
Brief Title: Ketamine for the Treatment for Alcohol Use Disorder in the ED
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: After months of screening, we screened 175 individuals, only 3 were eligible, 2 declined, and 1 was moved to a different floor before study activities were able to take place.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022P002550; 1R21AA030372-01A1 (NIH)
Record Dates: First submitted 2022-11-21; First posted 2022-12-22 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (Experimental): This arm will receive ketamine (n=25)
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): This arm will receive the saline placebo (n=25)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketamine — The intervention will consist of a single infusion of ketamine in the ED at a dose of 0.8mg/kg over 40 minutes.
  Arms: Ketamine
Drug: Saline — The placebo will be a 0.9% saline solution administered over 40 minutes.
  Arms: Placebo

SUMMARY:
The investigators' approach is to conduct a pilot double-blind, placebo-controlled randomized clinical trial with individuals with alcohol use disorder (AUD) seeking inpatient alcohol detoxification in the emergency department (ED) to receive either intravenous ketamine or saline placebo. The primary aim is to evaluate the intervention's safety. The secondary aim is to evaluate the preliminary efficacy of alcohol-related outcomes.

DETAILED DESCRIPTION:
This is a pilot double-blind, placebo-controlled randomized clinical trial of 50 individuals with alcohol use disorder (AUD) presenting to the emergency department (ED) seeking inpatient detoxification to receive either a single infusion of ketamine 0.8mg/kg (n=25) or saline placebo (n=25). The study will be conducted at Brigham and Women's Faulkner Hospital (BWF), an urban, 171-bed hospital located in Boston, MA, and a major teaching hospital for Harvard Medical School (HMS). Participants will be randomized in a double-blind fashion to receive either ketamine or saline placebo in the ED. All participants will receive the institution's standard treatment, which includes detoxification, intensive psychosocial support, and referral to outpatient treatment. The intervention (ketamine) will consist of a single infusion of ketamine in the ED at a dose of 0.8mg/kg over 40 minutes, and the placebo will be a 0.9% saline solution also administered over 40 minutes. To determine the safety of administering ketamine the investigators will measure the incidence of severe adverse events (AE), defined as either hypertensive urgency (systolic blood pressure>180mmHg or diastolic blood pressure>110mmHg) or tachycardia (heart rate>130bpm). The investigators will also assess side effects, alcohol withdrawal, and craving for alcohol and ketamine. To determine the preliminary efficacy of ketamine on alcohol-related outcomes, the investigators will measure the proportion of abstinent days during the follow-up assessed using Timeline Follow-Back (TLFB). The investigators will also measure days to relapse, the proportion of heavy drinking days, engagement with addiction treatment, urine ketamine, and alcohol biomarkers (urine ethylglucuronide and serum phosphatidylethanol) at 28-days. The investigators hypothesize that results will show adequate safety and that those receiving ketamine, compared to placebo, will not experience more side effects, worse withdrawal, or greater alcohol or ketamine craving. The investigators also hypothesize that those receiving ketamine will report better drinking outcomes compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults aged 18 and above
* Diagnosed with DSM5 alcohol use disorder, severe
* Admitted to BWF inpatient withdrawal management unit (Addiction Recovery Program)

Exclusion Criteria:

* Any psychotic disorder, bipolar disorder, active suicidality or homicidality
* Inability to perform consent due to impaired mental status
* Clinical Institute Withdrawal Assessment (CIWA) score > 20 at any point in the ED
* Alcohol withdrawal seizure prior to or during the ED visit
* Systolic blood pressure persistently elevated above 180mmHg, or heart rate >130bmp, in the ED
* History of hypersensitivity to ketamine, or experience of emergence reaction
* History of any illicit or recreational use of ketamine
* Receipt of ketamine treatment for depression in the past 3 months
* History of DSM5 hallucinogen use disorder, intracranial mass or bleed, porphyria, thyrotoxicosis, seizure disorder other than from alcohol withdrawal, liver cirrhosis, renal failure, obstructive lung disease, or sleep apnea
* History within 6 months of head trauma, stroke, or myocardial infarction
* Liver dysfunction with LFTs >3x upper normal limit
* Current use of medications with known drug-drug interactions with ketamine (i.e., St. John's Wort, theophylline, opioid analgesics, CNS depressants other than benzodiazepines or phenobarbital)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Safety of administering ketamine in the emergency department (ED) for alcohol use disorder (AUD) patients seeking detoxification | Outcomes will be assessed throughout the inpatient admission, on average 3-5 days and throughout duration of study.
  The incidence of severe adverse events (AE), defined as either hypertensive urgency (systolic blood pressure>180mmHg or diastolic blood pressure>110mmHg) or tachycardia (heart rate>130bpm). Adequate safety will be defined as <10% of participants experiencing severe AEs.

SECONDARY OUTCOMES:
Dissociative effects | Baseline, daily during inpatient (average 3-5 days), 28 days, and 3, 6, and 12 months after inpatient treatment.
  Clinician-Administered Dissociative States Scale (CADSS)
Alcohol withdrawal | Assessed during the inpatient admission, on average 3-5 days.
  Clinical Institute Withdrawal Assessment (CIWA)
Craving for alcohol | Assessed during the inpatient admission, on average 3-5 days; 7, 14, 28 days and 3, 6, and 12 months after treatment
  Alcohol craving questionnaire
Craving for ketamine | Assessed during the inpatient admission, on average 3-5 days; 7, 14, 28 days and 3, 6, and 12 months after treatment
  Visual analog scale
Cue-induced craving | Assessed during the inpatient admission, on average 3-5 days; 28 days after treatment
  Visual analog scale will be used to rate the craving following a standardized protocol used to assess cue reactivity. The cue exposure procedure will end with a standardized relaxation exercise.
Preliminary efficacy of ketamine on days to alcohol relapse | 7, 14, 28 days and 3, 6, and 12 months after treatment
  Days to relapse will be measured by using the Timeline Follow-Back (TLFB).
Preliminary efficacy of ketamine on proportion heavy drinking days | 7, 14, 28 days and 3, 6, and 12 months after treatment
  The proportion of heavy drinking days will be measured by using the Timeline Follow-Back (TLFB).
Preliminary efficacy of ketamine on engagement with addiction treatment | Measured at baseline, 28 days, and 3, 6, and 12 months post treatment.
  The Alcoholic Anonymous Affiliation Scale (AAAS) will be used to measure engagement with addiction treatment. This is a 9-item scale to measure the degree of involvement with Alcoholics Anonymous.
Ketamine in Urine | At baseline and 28 days after treatment
  Urine drug screen that includes ketamine will be assessed.
Urine ethylglucuronide | At baseline and at 28 days after treatment
  Urine ethylglucuronide (EtG) will be obtained
Phosphatidylethanol (PEth) | At baseline and at 28 days after treatment
  Serum phosphatidylethanol (PEth)
Behavior Change Mechanisms | Once during inpatient treatment and at 28 days after treatment
  Mechanisms of behavior change will be measured using tools from the Science of Behavior Change Measures.
Anxiety | At baseline, each day during treatment (3-5 Days on average), 7, 14, 28 days and 3, 6, and 12 months after treatment
  We will assess anxiety levels utilizing a 7-item scale (Generalized Anxiety Disorder - 7 (GAD-7))
Depression | At baseline, each day during treatment (3-5 Days on average), 7, 14, 28 days and 3, 6, and 12 months after treatment
  We will assess depression levels utilizing a 9-item scale (Patient Health Questionnaire-9 (PHQ-9))
Suicidal Ideation | At baseline, each day during treatment (3-5 Days on average), 7, 14, 28 days and 3, 6, and 12 months after treatment
  Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess suicidal Ideation
Post Traumatic Stress | Once during treatment
  A patient self-report tool developed to examine PTSD symptoms in general medical settings (Abbreviated PTSD Checklist - Civilian Version)
Study Drug Side Effects | At baseline, each day during treatment (3-5 Days on average), 7, 14, 28 days and 3, 6, and 12 months after treatment
  We will use Patient Rated Inventory of Side Effects (PRISE) to qualify side effects in the following domains: gastrointestinal, heart, skin, nervous system, eyes/ears, genital/urinary, sleep, sexual functioning, and other. Each domain has multiple symptoms which can be endorsed. For each domain the patient rates whether the symptoms are tolerable or distressing.
Spirituality | Baseline, once during treatment, and at 28 days post treatment.
  We will use a 23-item measure to assess spirituality (Spirituality Scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Faulkner Hospital, Boston, Massachusetts, United States